CLINICAL TRIAL: NCT03259893
Title: Boston Medical Center Secondary Prevention of Atrial Fibrillation Randomized Pilot Study
Brief Title: Secondary Prevention of Atrial Fibrilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initially suspended due to COVID-19 policies, it will not be possible to restart.
Sponsor: Boston Medical Center (Other)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-36040; H-36040 (Other Grant/Funding Number: Boston Medical Center through CTSI)
Record Dates: First submitted 2017-07-04; First posted 2017-08-24 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-05

CONDITIONS: Atrial Fibrillation; Risk Factors; Risk Reduction Behavior
Keywords: Proctor Conceptual Model of Implementation Research; Prevention; Safety net hospital; Diverse inner city patients
MeSH Terms: conditions — Atrial Fibrillation; Risk Reduction Behavior | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of care group 1 (Active Comparator): Participants randomized to the standard of care group will receive guideline-directed medical therapy according to clinical standard practice at Boston Medical Center. Each participant will receive an AliveCor mobile ECG cardiac monitor which is capable of providing real-time heart telemetry using a smart phone.
  Interventions: Other: AliveCor mobile ECG cardiac monitor; Other: Standard of care
- Intervention group 2 (Experimental): The intervention group will receive the AF program which include a bundle of sub-interventions that target specific AF risk factors including hypertension, obesity, physical inactivity, sleep hygiene, and smoking. Each participant will receive an AliveCor mobile ECG cardiac monitor which is capable of providing real-time heart telemetry using a smart phone.
  Interventions: Other: AliveCor mobile ECG cardiac monitor; Behavioral: AF Program

INTERVENTIONS:
Other: AliveCor mobile ECG cardiac monitor — AliveCor mobile ECG cardiac monitor is capable of providing real-time heart telemetry using a smart phone. Participants will be instructed to transmit rhythm data twice weekly and during symptomatic AF.
Behavioral: AF Program — The AF program includes a bundle of sub-interventions that target specific AF risk factors including hypertension, obesity, physical inactivity, sleep hygiene, and smoking. Participants randomized to the intervention group 2 will undergo counseling by the nurse and guided through the structured, goal-directed AF program. Each participant will receive an AliveCor cardiac monitor which is capable of providing real-time heart telemetry using a smart phone.
  Arms: Intervention group 2
Other: Standard of care — Guideline-directed medical therapy according to clinical standard practice at Boston Medical Center.
  Arms: Standard of care group 1

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia affecting over 3 million Americans and about 33.5 million individuals globally. The lifetime risk of developing AF is 1 in 4 for adults over age 40 years. AF is associated with a major medical and socioeconomic burden including high cost, increased risk of stroke, heart failure, dementia, myocardial infarction, and death. Numerous studies have demonstrated that modifiable risk factors including hypertension, obesity, sleep apnea, diabetes, and sedentary lifestyle predict the development of AF.

Recent studies have reported that secondary prevention interventions through aggressive risk factor modification can reduce the burden of AF. Structured, physician and nursing-led interdisciplinary AF programs have been shown to improve patient adherence to guideline recommendations and improve long term prognosis. Previous data, however, are derived mainly from white European and Australian cohorts and it is unclear whether such interventions can be effectively implemented in a racially diverse, safety net hospital in the U.S.

This study is a randomized hybrid implementation-effectiveness study designed to investigate feasibility and effectiveness of an evidence-based innovative AF program, focusing on risk factor modification and AF education in a racially mixed population receiving care in a safety net hospital.

DETAILED DESCRIPTION:
The proposed study is designed as a Hybrid Type 3 effectiveness-implementation study. This study design will enable the investigators to primarily focus on core implementation outcomes while also assessing the effectiveness of the intervention on clinical outcomes. Since this is a Type 3 Hybrid trial, there are both effectiveness and implementation evaluation components, but the primary focus is on the implementation outcomes of feasibility, acceptability, adoption, and appropriateness. The specific aims, data collection, and analytic plans are grounded in the Proctor Conceptual Model of Implementation Research that posits improvements in outcomes are dependent not only on the evidence-based interventions that are implemented but on the implementation strategies used to implement those interventions. The model distinguishes between the intervention strategy (evidence-based practice), different types of implementation strategies (system environment, organizational, group/learning, supervision, individual providers/consumers), and three levels of outcomes (implementation, service, and client). The appropriate outcome measures in each category (implementation, service, client) depend upon the specific evidence-based practice and local context.

AF patients with a BMI of ≥ 27 kg/m2, who are referred to outpatient cardiology clinic, inpatient cardiology service, or cardiology consult service at Boston Medical Center (BMC) will be screened until 50 participants are enrolled. Eligible participants will undergo 1:1 randomization to standard of care (SoC -group 1) or to the interdisciplinary AF program (intervention- group 2). Randomization will be performed using a computer randomizer algorithm with 5 blocks of 6 and 5 blocks of 4 in random order for a total of 50 participants. The rational for the randomization design is primarily for the purpose of feasibility and to establish effect sizes and guide the design of the future trial.

All patients will be enrolled for a total duration of six months. Outcomes will be measured via 30-minute individual interviews at the end of 6-months. The implementation and service outcomes will be examined including acceptability, appropriateness, adoption, feasibility, and patient centeredness, as well as the client outcomes of satisfaction, function and symptomatology. Data will be collected using both quantitative and qualitative data methods to determine which aspects of the program achieved good patient adherence and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of paroxysmal AF (based on 12-lead electrocardiogram or event monitor showing AF).
* Body mass index of greater than 27 kg/m2
* Eligibility to participate in cardiac rehabilitation with negative exercise stress test within 6 months.

Exclusion Criteria:

* Permanent AF.
* Undergone catheter ablation of AF in past 6 months.
* Class I or Class III anti-arrhythmic drugs at the time of enrollment
* Unable to participate in cardiac rehabilitation.
* Prognosis of less than 1-year.
* Do not own a smart phone.
* Unable to operate (transmit data) their smart phone.
* Are not fluent in English or Spanish.
* Unable to read in English or Spanish.
* Not able to provide informed consent.
* Women who are pregnant.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of the AF program | 6 months
  Quantitative measure of willingness to enroll and attend nutrition clinic, cardiac rehabilitation clinic, and frequency of use of Alivecor device, smart Scale, Fitbit device will be aggregated to generate a single feasibility score to determine overall feasibility of the AF program.
  The feasibility score will be generated by the following formula:
  = 100 * average of { (actual nutrition clinic attendance/ expected nutrition clinic attendance) + (actual cardiac rehab clinic attendance/ expected cardiac rehab clinic attendance) + (actual use of smart phone enabled devices/expected use of smart phone enabled devices)}
  A feasibility score closer to 100% indicates good feasibility.

SECONDARY OUTCOMES:
Acceptability of the AF program | 6 months
  Data from qualitative interviews will be coded using a process analytic framework and inductive logic to create a set of conceptual categories using the Constant Comparative Method and used to assess patient-centeredness and satisfaction which will reflect acceptability of the AF program.
Most acceptable individual component of the AF program | 6 months
  Data from qualitative interviews will be coded using a process analytic framework and inductive logic to create a set of conceptual categories using the Constant Comparative Method and used to compare the acceptability of individual component of AF programs including nutrition clinic, cardiac rehabilitation clinic, smoking cessation clinic, smart phone enable health devices.
Most adopted individual component of the AF program | 6 months
  Quantitative measure of (actual clinic attendance or use of smart phone enable devices) / (expected clinic attendance or use of smart phone enable devices) will be compared for the various components of the AF program including nutrition clinic, cardiac rehabilitation clinic, smoking cessation clinic, Alivecor device, Fitbit device, smart blood pressure monitor, and smart scale. The individual component with the highest % attendance or use will be considered to be the most adopted individual component of the AF program.
Burden of atrial fibrillation | Twice weekly for 6 months
  Quantitative measure of telemetry data from Alivecor devices, participants will be instructed to transmit telemetry data twice weekly and during symptomatic AF episodes. Telemetry data showing AF will be used to determine number of AF episodes in each participant over time.
Atrial fibrillation symptoms | 6 months
  quantitative measure of telemetry data from Alivecor devices and qualitative measures using The Atrial Fibrillation Effect on QualiTy of Life (AFEQT) questionnaire is a 20 question, 7 point Likert scale (1-7) instrument that takes about 5 minutes to complete and evaluates Health Related Quality of Life across 3 domains- symptoms (4 questions), daily activities (8 questions), and treatment concerns (6 questions). The range of scores are 20-140, lower scores are favorable.
Atrial fibrillation literacy | 6 months
  AF Knowledge Questionnaire is a 34 question instrument that takes about 10 minutes to complete. It is a modified version of the Jessa Atrial fibrillation Knowledge Questionnaire (JAKQ) and contains questions about AF in general and about oral anticoagulation therapy.
Atrial Fibrillation Effect on Quality of Life | 6 months
  The Atrial Fibrillation Effect on QualiTy of Life (AFEQT) questionnaire is a 20 question, 7 point Likert scale (1-7) instrument that takes about 5 minutes to complete and evaluates Health Related Quality of Life across 3 domains- symptoms (4 questions), daily activities (8 questions), and treatment concerns (6 questions). The range of scores are 20-140, lower scores are favorable.
Hospitalization for atrial fibrillation | 6 months
  quantitative measure of number of hospitalization for atrial fibrillation or outcome attributed to atrial fibrillation

OTHER OUTCOMES:
Weight loss | 6 months
  Quantitative measure of total weight loss over the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Helm, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No